CLINICAL TRIAL: NCT00455299
Title: Randomized Controlled National Multicenter Study for Evaluation of Two Different Ways of Fixation of Mesh-implants and Differences With or Without Approximation of Herniadefects at Laparoscopic Operation for Incisional and Ventral Hernia
Brief Title: LVHR Multicenter Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Tyco Healthcare Group (Industry)
Responsible Party: Principal Investigator, Jan Lambrecht, MD, Oslo University Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: S-06466b
Record Dates: First submitted 2007-04-02; First posted 2007-04-03 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Ventral and Ventral Insicional Hernia
Keywords: Laparoscopy, ventral, hernia, repair, surgery
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- a (Active Comparator): a: suture anchoring + tackers and approximation of defect
  Interventions: Procedure: Laparoscopic ventral hernia repair
- b (Active Comparator): b: suture anchoring + tackers without approximation of defect
  Interventions: Procedure: Laparoscopic ventral hernia repair
- c (Active Comparator): c: only tacker fixation and approximation of defect
  Interventions: Procedure: Laparoscopic ventral hernia repair
- d (Active Comparator): d: only tacker fixation without approximation of defect
  Interventions: Procedure: Laparoscopic ventral hernia repair

INTERVENTIONS:
Procedure: Laparoscopic ventral hernia repair

SUMMARY:
The study aims to prove differences or equalities in outcome for patients operated with laparoscopic ventral hernia repair with different methods of fixation of mesh and with or without approximation of defect prior to meshfixation.

DETAILED DESCRIPTION:
Patients are randomized to 4 groups: non-absorbable suture fixation and hernia approximation, double crown mesh fixation with titanium spiral tacks with hernia approximation and the same fixations without hernia approximation.

Primary endpoint is recurrence. Secondary endpoints are operating time, adhesion score, mode of entering abdominal cavity, time to recovery, pain durance, seroma formation, aesthetic result (protrusion), organ traumatization infection. Endpoints are correlated to hernia size, body mass index, previous recurrence, age, concurrent illness. Patients are followed 3 years after operation with clinical examination.

300 patients are planned included in primary study. A subgroup of organ transplanted patients is evaluated in a separate study with identical criteria for inclusion.

ELIGIBILITY:
Inclusion Criteria:

* secondary or primary ventral hernia

Exclusion Criteria:

* Loss of domain, Giant hernia with need of abdominal plastic operation, ASA score above 3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2007-03; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Operating time | 30-180 min
Adhesion score
Mode of entering abdominal cavity
Pain durance | 8 weeks
Seroma formation
Aesthetic result (protrusion) | 3 years
Infection | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jan Lambrecht, MD, Principal Investigator — Oslo University Hospital
Locations (2):
- Norway (2):
  - SIHF Gjøvik, Gjøvik
  - Ullevål University Hospital, Oslo

REFERENCES:
- [Derived] Lambrecht JR, Vaktskjold A, Trondsen E, Oyen OM, Reiertsen O. Laparoscopic ventral hernia repair: outcomes in primary versus incisional hernias: no effect of defect closure. Hernia. 2015 Jun;19(3):479-86. doi: 10.1007/s10029-015-1345-x. Epub 2015 Feb 7. PMID 25663605
- [Derived] Lambrecht JR, Skauby M, Trondsen E, Vaktskjold A, Oyen OM. Laparoscopic repair of incisional hernia in solid organ-transplanted patients: the method of choice? Transpl Int. 2014 Jul;27(7):712-20. doi: 10.1111/tri.12327. Epub 2014 May 9. PMID 24684675